CLINICAL TRIAL: NCT04709679
Title: Clinical Outcome of Varying Doses of Micropulse TransScleral CycloPhotocoagulation Laser in Patients With Glaucoma.
Brief Title: Laser Dosage in MicroPulse TransScleral CycloPhotocoagulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dose was not therapeudic
Sponsor: State University of New York at Buffalo (Other)
Collaborators: IRIDEX Corporation (Unknown)
Responsible Party: Principal Investigator, Sandra Sieminski, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003149
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Glaucoma
Keywords: MP-TSCPC; Laser Duration; Laser Dwell time; Laser Power
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Constant dwell time but varying power and duration (Experimental): The laser dwell time will be constant but the laser power and duration will be varied for patients
  Interventions: Procedure: MicroPulse TransScleral CycloPhotoCoagulation
- Constant power but varying dwell time and duration (Experimental): The laser power will be constant but the laser dwell time and duration will be varied for patients
  Interventions: Procedure: MicroPulse TransScleral CycloPhotoCoagulation
- Constant duration but varying dwell time and power (Experimental): The laser duration will be constant but the laser dwell time and power will be varied for patients
  Interventions: Procedure: MicroPulse TransScleral CycloPhotoCoagulation

INTERVENTIONS:
Procedure: MicroPulse TransScleral CycloPhotoCoagulation — A laser power of 2000- 2500 mW, a laser duration time of 50 to 80 sec per hemifield and varying da number of sweeps per hemifield 3, 4 or 5 will be randomized between patients

SUMMARY:
This is a prospective study to evaluate the clinical outcome of varying doses of Micropulse TransScleral CycloPhotocoagulation (MP-TSCPC) laser in patients with glaucoma. The study will assess documented complication rates, changes in visual acuity after the procedure, changes in intraocular pressures and medication drop usage, and need for subsequent treatments (including further laser or surgery).

DETAILED DESCRIPTION:
Glaucoma is a condition where an increase in the accumulation of aqueous humor inside the anterior chamber of the eye results in raised intraocular pressure (IOP), visual field defects and cupping of optic disc. Typically, patients who have glaucoma are treated with topical medications or incisional surgery to lower the IOP. Micropulse transscleral cyclophotocoagulation (MP-TSCPC) is a non-incisional laser surgery used in the treatment of glaucoma. MP-TSCPC powered by the Cyclo G6 (Iridex Corporation, Mountain View, CA, USA) causes mild thermal damage to the ciliary body (gland that produces aqueous fluid in the eye), which, in turn, causes a decrease in intraocular pressure. MP-TSCPC is a variation of a longstanding older treatment for glaucoma, traditional diode TSCPC, which caused a significant amount of tissue damage and therefore was reserved for the treatment of end stage glaucoma.

The micropulse laser application includes an on-off cycle. In an on cycle, the micropulse probe administers a short pulse of laser energy followed by an off cycle which is a rest period for the tissue to cool off before the next on-off cycle begins. This corresponds to 0.5 ms duration of "on-time" and 1.1 ms interval of "off-time" during the laser application. This on-off cycle allows for the laser to treat the affected area without evidence of tissue damage, as opposed to the traditional diode TSCPC. Because only 31.3% of the total laser energy is applied to the ciliary body, there is a less tissue damage, less post-operative inflammation, and decreased complication rates. Therefore, MP-TSCPC is currently being utilized for milder cases of glaucoma, and in patients with viable vision. The laser probe is usually applied perpendicular to the limbus in a continuous sweeping motion, for an average of 10 seconds of sweeping time per hemifield, referred to as "dwell time". Therefore, the three parameters that can be varied in the treatment with MP-TSCPC are total laser duration (seconds), laser power (mW) and dwell time (seconds/hemifield).

Most of the studies used a laser power of 2000 - 2500 mW. The laser duration also has varied between studies. A duration time of 50 to 180 sec per hemisphere was used in different studies. Most studies have utilized a dwell time of 10 seconds per hemifield, and one cited an application of a "stop and go" method, applying the laser in discrete spots at 10 seconds each.

In all of the prior studies, despite the variable applications of power, dwell time, and duration, there have been similar rates of complications such as vision loss, macular edema, and hypotony. Generally, the laser duration is tailor-made and is adjusted based on the iris color and severity of glaucoma. However, there is a gap in knowledge on systematic comparison of different doses of MP-TSCPC for a safe and effective treatment of glaucoma. This study will systematically evaluate the clinical outcome of glaucoma surgery based on a logical variation of MP-TSCPC laser dosing parameters.

ELIGIBILITY:
Inclusion Criteria:

* Decision to treat by MP-TSCPC Laser
* Patients diagnosed with Glaucoma
* Patients aged 18 years old and above
* Glaucoma that is inadequately controlled on medical therapy
* Patients with primary open angle glaucoma with or without previously failed trabeculectomy or other aqueous drainage surgical procedures

Exclusion Criteria:

* Patients age less than 18 years
* Patients unable or unwilling to provide informed consent to participate in the study
* Patients potentially unavailable for follow up visits
* Patients with significant scleral thinning
* Patients with ocular infection, inflammation or intraocular surgery in the study eye 2 months prior to enrollment in the study
* Albino patients that have no iris pigmentation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Changes in intraocular pressure measurements between baseline and postoperative followup visits | 2years
  Baseline (pre-operative condition) and post operative intraocular pressure will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.

SECONDARY OUTCOMES:
Changes in visual acuity measurements measured using a Snellen Vision Chart between baseline and postoperative followup visits | 2 years
  Baseline (pre-operative condition) and post operative visual acuity will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.
Changes in number of medications between baseline and postoperative followup visits | 2 years
  Baseline (pre-operative condition) and post operative number of medications list will be measured on Day1, Week1, Months 1, 3, 6, 12, 18 and 24.
Rate of post surgical complications | 2 years
  Rate of post surgical complications such as Hypotony, Corneal Edema, Hyphema, Iritis, Vitreous Hemorrhage and Cystoid Macular Edema.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra F Sieminski, MD, Principal Investigator — Ross Eye Institute
Locations (1):
- The Ira G. Ross Eye Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No